CLINICAL TRIAL: NCT06036940
Title: COMPARISON OF 3 DIFFERENT METHODS FOR REDUCING THE LEVEL OF PERIOPERATIVE ANXIETY IN CHILDREN AGED 4-7: A RANDOMIZED CONTROLLED STUDY
Brief Title: Perioperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Tülin YILDIZ, Prof. Dr., Namik Kemal University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TYILDIZ
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Nurse's Role
Keywords: Anxiety; child sick; surgical nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Control Group (No Intervention): The children in the first control group were given pre-operative patient education by the service nurse.
- Second Experimental Group (Experimental): The children in the second experimental group were given pre-operative patient education by the service nurse, also patient visits were provided by the operating room nurse and the operating room environment was explained through play.
  Interventions: Other: Preoperative patient education given with three different methods
- Third Experimental Group (Experimental): The children in the third experimental group were given pre-operative patient education by the service nurse, and then the mother's voice recording was played until they went to the operating room.
  Interventions: Other: Preoperative patient education given with three different methods

INTERVENTIONS:
Other: Preoperative patient education given with three different methods — To determine the effect of preoperative patient education given by three different methods on the level of perioperative anxiety in children aged 4-7 years.
  Arms: Second Experimental Group; Third Experimental Group

SUMMARY:
The study was conducted to evaluate the effect of preoperative patient education given by three different methods on the level of perioperative anxiety in children aged 4-7 years. The research was carried out between 1 June - 31 November 2021 at Tekirdag Namık Kemal University Health Practice and Research Center, Department of Pediatric Surgery. A total of 66 patients, 22 patients in each group, who met the inclusion criteria and were included in the stratified randomization method, were included in the planned quasi-experimental study. Research data were obtained by using the "Patient Diagnosis Form" and the "Anxiety Scale in Preschool Children" administered before and after the surgery.

DETAILED DESCRIPTION:
Pre-operative patient education was given to the children in the first experimental group by the service nurse. The children in the second experimental group were given pre-operative patient education by the service nurse, in addition, patient visits were provided by the operating room nurse and the operating room environment was explained through play. The children in the third experimental group were given pre-operative patient education by the service nurse, after which they listened to the mother's voice recording and loving words until they went to the operating room. It was determined that 69.7% of the mothers of the children participating in the study were 30 years and older, 81.8% were married, 37.9% were undergraduate graduates, and 51.5% were unemployed. The general anxiety disorder levels of those who had no previous surgery experience were found significantly higher than those who had previous surgery experience (p<0.05). In terms of affecting the anxiety level, there was a significant difference between the preoperative methods (p<0.05). It was determined that the education given by both the service nurse and the operating room nurse together was more effective than other methods in reducing the anxiety levels of children, and there was a statistically significant difference between them. (p<0.05)

ELIGIBILITY:
Inclusion Criteria:

* Planned elective surgery related to pediatric surgery,
* Having no problems in communicating,
* Volunteer to participate in the research
* Children aged 4-7 years

Exclusion Criteria:

* Children scheduled for emergency surgery

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Patient Diagnosis Form | 5 month
  This section consists of a total of 11 questions prepared by the researcher in the light of the literature, including the introductory characteristics of patients and mothers, their previous surgical experience and their expectations from nurses.

SECONDARY OUTCOMES:
Anxiety Scale in Preschool Children | 5 month
  Anxiety Scale for Preschool Children consists of a 5-point Likert scale. It is scored from 0 (not at all true), 1 (rarely true), 2 (sometimes true), 3 (quite true), 4 (very often true), from 0 to 4, and parents are expected to evaluate their children. The original scale measures 4 factors. These factors should consist of 4 sub-dimensions, social anxiety disorder, generalized anxiety disorder, separation anxiety disorder, and specific phobia. There are 29 items that are expected to be answered in total. Cronbach's Alpha values of the sub-dimensions range from .72 to .92.

CONTACTS AND LOCATIONS:
Overall Officials: Tülin YILDIZ, Prof. Dr., Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Suleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No